CLINICAL TRIAL: NCT01568372
Title: Efficacy of a Nurse Telephone Follow-up on Post-tonsillectomy Pain Management and Complications in Children: A Randomized Clinical Trial
Brief Title: Efficacy of a Nurse Telephone Follow-up on Pain Intensity After Removal of Tonsils in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Julie Paquette, Nurse Clinician Specialist, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Tonsils
Record Dates: First submitted 2012-03-26; First posted 2012-04-02 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Pain
Keywords: pediatric; tonsillectomy; pain management; nurse follow-up
MeSH Terms: conditions — Pain; Agnosia | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse telephone follow-up (Experimental): This group received a telephone follow-up by a nurse following discharge from the hospital and up until the 10th postoperative day, which is considered as the usual period of healing for a tonsillectomy
  Interventions: Other: Telephone follow-up
- Standard care group (No Intervention): This group received the standard care which consisted of an informative session before discharge and no follow-up once discharged home.

INTERVENTIONS:
Other: Telephone follow-up — The intervention group received a telephone follow-up by a nurse on the 1st, 3rd, 5th and 10th postoperative day.
  Other Names: Nursing interventions; Nursing follow-up
  Arms: Nurse telephone follow-up

SUMMARY:
The purpose of this study is to determine if a nurse telephone follow-up to parents of children who underwent a removal of their tonsils would be effective in reducing pain intensity, complications and resort to other healthcare services

DETAILED DESCRIPTION:
Tonsillectomy in children is a common elective day surgery. In the United States, 530 000 children under 15 years of age underwent a tonsillectomy in 2006. This minor surgery generates moderate to severe pain and many postoperative complications, both in the early postoperative phase and for at least 7 days. Patients are discharged home a few hours after tonsillectomy, and parents take over their child's care. But not all parents have the ability and knowledge required to adequately manage the pain and complications. This sub-optimal care situation has a significant impact on the child's convalescence and can lead to poor pain management, dehydration, poor rest and sleep quality, nausea, vomiting as well as an increase in the risk of secondary haemorrhage. Many interventions have been evaluated to improve pain management, such as education strategies for parents or children and tools to guide parents. However, none of these strategies have obtained significant results on children's pain intensity post-tonsillectomy.

A nurse telephone follow-up can significantly reduce pain intensity of adults who undergo ambulatory surgery. This intervention is defined as multiple telephone calls made to the patient by a nurse, after discharge, to provide information, and review discharge prescriptions and management of care by the patient himself or by a care-giver. Only a few studies have explored nurse telephone follow-up for children who underwent tonsillectomy. The design of these studies, including the time-periods chosen for data collection, were not properly determined to adequately evaluate the impact of the intervention on management of pain and prevention of postoperative complications. Thus, we planned to determine if a nurse telephone follow-up, made to parents following their child's tonsillectomy, would contribute to decrease pain intensity, incidence of postoperative complications and resort to other healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* Elective surgery for tonsillectomy
* Parents or children able to read, and understand French or English
* Family equipped with a phone at home
* Child discharged home after the surgery

Exclusion Criteria:

* Abused cases
* Children with a cognitive deficit
* Children suffering from chronic pain
* Child who had another surgical procedure within a month

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity scores on the 3rd day after surgery | Pain assessed on the 3rd postoperative day
  Mean pain intensity score on the 3rd postoperative day (POD)
Pain intensity scores on the 5th day after surgery | Pain assessed on the 5th postoperative day
  Mean pain intensity score on the 5th postoperative day (POD)
Pain intensity scores on the 10th day after surgery | Pain assessed on the 10th postoperative day
  Mean pain intensity score on the 10th postoperative day (POD)

SECONDARY OUTCOMES:
postoperative complications | Complications assessed on the following postoperative days: First day, 3rd day, 5th day and 10th day
  Assess complications and adverse events at each time points of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, PhD, Principal Investigator — Université de Montréal
Locations (1):
- CHU Ste.Justine's, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Paquette J, Le May S, Lachance Fiola J, Villeneuve E, Lapointe A, Bourgault P. A randomized clinical trial of a nurse telephone follow-up on paediatric tonsillectomy pain management and complications. J Adv Nurs. 2013 Sep;69(9):2054-65. doi: 10.1111/jan.12072. Epub 2013 Jan 13. PMID 23311981